# Clinical Evaluation of Genetron TERT PCR Kit in Glioma Patients

Study Document

NTC number: NCT05100602

Date: 02/01/2016

# Content

| 1 Background | 1 |
|----------------------------------------------------------------------|----|
| 2 Test Purpose | 3 |
| 3 Trial Design | 3 |
| 3.1 Overall Design of the Trial | 3 |
| 3.2 Test design and study method selection | 4 |
| 3.3 Study technology route | 5 |
| 3.4 Quality control method | 6 |
| 4 Evaluation method | 6 |
| 4.1 Evaluation method for reagents to be tested | 6 |
| 4.2 Evaluation method for nucleic acid sequence determination | 7 |
| 4.3 Evaluate the conformity between the kit and the reference method | 7 |
| 5 Statistical methods | 8 |
| 6 Duration of clinical trials and its reasons | 8 |
| 7 Inclusion criteria, exclusion criteria and rejection Criteria | 8 |
| 7.1 Inclusion criteria | 8 |
| 7.2 Exclusion criteria | 8 |
| 7.3 Rejection Criteria | 9 |
| 8 Provisions for amendments to clinical trial protocols | 9 |
| 9 Ethical issues and explanations of clinical trials | 9 |
| 10 Data processing and record keeping | 10 |

### 1 Background

Glioma is the most common primary intracranial tumor. According to the ranking of tumor mortality published by the World Health Organization in 1998, malignant glioma is the second leading cause of death among tumor patients under 34 years old and the third among patients between 35 and 54 years old. In the past 30 years, the incidence of primary malignant brain tumors has been increasing year by year, with an annual growth rate of about 1.2%, especially in the elderly population. At present, WHO mainly relies on morphology for tumor classification and typing (Table 1). However, due to the heterogeneity of glioma and the subjective influence of pathologists, this method is highly subjective and one-sided. There is ample evidence that gliomas with the same or similar tissue characteristics can have different molecular genetic backgrounds. Molecular pathological classification based on tumor genetics can provide accurate and objective genetic information for tumor diagnosis, to help doctors understand the characteristics of each patient's tumor from a new perspective of molecular biology, so as to make more targeted treatment and rehabilitation programs.

Table 1 WHO pathological classification and classification of glioma

| Tissue<br>types | Class | Common subtype |
|---|---|---|
| Glioma of the brain | Class I | Pilocytic astrocytoma, subependymal giant cell astrocytoma embryona dysplasia of neuroepithelial tumors |
| | Class II | Diffuse astrocytoma, mixed oligoastrocytomas, oligodendroglioma, pleomorphic xanthoastrocytoma, hairy myxoid astrocytoma |
| | Class III | Anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic oligoastrocytomas |
| | Class IV | Primary and secondary glioblastoma |

Telomerase is a kind of nucleic acid protein complex composed of two subunits of Telomerase RNA and Telomerase reverse transcriptase (TERT), which plays a key role in the maintenance of Telomerase length. TERT gene promoter mutation is one of the important mechanisms of abnormal telomerase expression in tumors. The most common mutation sites in glioma are C228T and C250T, which usually occur independently of each other. It has been proved that the mutation can enhance the transcriptional activity of TERT promoter and is a key cause of tumor occurrence and development.

Recently, important studies have found that TERT mutations are commonly high in primary glioblastoma and oligodendroglioma, but low in astrocytomas. The researchers also detected the TERT gene promoter and IDH gene together. According to the mutation status of the two genes simultaneously or independently, the most typical subtypes of glioma could be further distinguished significantly: TERT mutations were found in 74.2% of primary glioblastoma patients among 473 adult gliomas, but only in 18.2% of class II-III astrocytomas. In contrast, IDH mutations were observed in 78.4% of class II-III astrocytomas, but were infrequent in primary glioblastoma. TERT promoter mutations co-occurred with IDH mutations in 79% of oligodendrogliomas (Figure 1). Subsequently, several important multi-center, large-scale clinical trials fully supported this conclusion.



Figure 1: The distribution of TERT gene promoter and IDH1/2 gene mutations in 473 adult glioma patients.

The gene mutations are indicated by color, red indicating the TERT gene promoter mutation, green indicating the IDH1/2 gene mutation, and light gray indicating that neither gene has mutation.

Therefore, for adult glioblastoma class III-IV patients, if TERT mutations is present alone, primary glioblastoma may be indicated, if IdH1/2 mutation is present alone, astrocytoma may be indicated, and if TERT and IDH1/2 mutations are present at the same time, oligodendroglioma may be indicated. These findings provide a unique diagnostic basis for promoting accurate classification of brain cancer.

The standard method for clinical detection of common gene promoter mutations is nucleic acid sequence determination, but this method is not sensitive enough, result judgment is time-consuming and laborious, and the operation process is complex, so this technology is difficult to be widely applied in clinical practice.

The kit to be tested was developed by Genetron Health (Beijing) Co., Ltd. It is mainly used for the detection of TERT gene promoter mutation in glioma patient cells. The tested product series of the kit is prepared in a clean production workshop that meets the requirements of the "Detailed Rules for the Production of In Vitro Diagnostic Reagents", and passed the self-test.

At present, there is no similar product on the market in China, so no similar kit can be used as a clinical trial control. The gold standard method for detecting common gene mutations is nucleic acid sequencing. In order to evaluate the clinical safety and effectiveness of this product, this clinical trial uses the qualified product provided by the manufacturer to retrospectively examine the tissue biopsy samples confirmed by pathology. The pathological types include gliomas, other brain tumors, and normal brain tissues, and the results of the nucleic acid sequence determination of the corresponding samples are used as controls for comparison.

# 2 Test Purpose

By using this product to detect the TERT gene promoter mutation in the cancer cells of glioma patients and comparing with the gene sequencing results, the safety and effectiveness of this product are confirmed and evaluated in combination with clinicopathological grading.

# 3 Trial Design

#### 3.1 Overall Design of the Trial

This study followed the principle of synchronous blind method. Enrolled cases were coded and compared with the nucleic acid sequence determination of the control method (gold standard). Results were determined independently according to the critical value or interpretation requirements provided by each method, and relevant statistics were conducted. Combined with the results of clinicopathological classification, the incidence of C228T and C250T mutations in different subtypes of TERT gene promoters was calculated to evaluate the clinical application performance for clinical research kits.

The total number of samples for clinical research should be no less than 1,000 cases, and clinical trials should be carried out in no less than 3 (including 3) provincial health care institutions or specialized hospitals to ensure that the results are statistically significant. All samples should have corresponding basic clinical information, including: patient visiting No. / medical record number/specimen number, age, sex, pathological diagnosis result, etc.

#### 3.2 Test design and study method selection

#### 3.2.1 Sample collection

Tissue sections fixed in neutral formaldehyde and embedded in paraffin were detected.

#### 3.2.2 Sample data

- (1) Sample information
  - A) Patient visiting No. / medical record No. / specimen No., age, sex, and pathological diagnosis result
  - B) HE staining results of samples, indicating tumor area.
- (2) Pathological examination confirmed glioma, other brain tumors or normal tissues.
- (3) Number of samples: each sample contains 10 slices with a thickness of 10μm, and the tumor content is not less than 50%.

#### 3.2.3 Sample storage

FFPE samples should be stored at room temperature.

#### 3.2.4 Kit source:

- (1) The kits were provided by Genetron Health (Beijing) Co., Ltd.
- (2) Test instrument: BIO-RAD: CFX96 Real-Time PCR Detection System or LIFE: 7500 Fast Dx Real Time PCR Instrument.

#### 3.2.5 Reference method

Sanger sequencing was used as the control method. Sequencing fragments cover the target nucleic acid segments, sites and corresponding types amplified by the assessment reagent. After the sequencing reaction is over, submit a representative sample sequencing map and result analysis data.

#### 3.2.6 Testing process

The test samples were tested in strict accordance with the kit operation instructions.

#### 3.3 Study technology route



#### 3.4 Quality control method

- (1) The clinical verification institutions are all three-level medical institutions above the provincial level with the ability to conduct the clinical research technology and equipment to ensure the quality of clinical diagnosis.
- (2) Each clinical trial institution has 1 project director, and 1 to 3 fixed project members. Strictly follow the requirements of the clinical trial protocol. The reporting institution appoints 1 inspector to monitor and cooperate with the team leader institution and the trail institution at any time. The technical personnel of the team leader institution keep close contact with each trail center at any time.
- (3) The test kit detection and reference method detection are carried out in accordance with the blind method.
- (4) Hospital laboratories participating in clinical trials should establish standard operating procedures and quality control procedures for experimental observation indicators. The test report must be complete, which must include date, test items, test results and their normal range. The person concerned should sign. Each test is set up control, and strictly in accordance with the requirements of the manual.
- (5) Training: Before the start of the experiment, conduct protocol training for all personnel participating in the experiment, and conduct training and assessment for clinical research staff, so that clinical trial personnel able to quickly become familiar with and master the fluorescence PCR technology and the applicable instruments, operating methods, and technical performance etc. of the kit.
- (6) This protocol has been determined through repeated communication and research between the experimental institution and the clinical institution, and must be strictly implemented. Any changes in the plan must be approved by the team leader (master) institution.

#### 4 Evaluation method

#### 4.1 Evaluation method for reagents to be tested

 The Ct value of FAM channel of positive control substance was ≤18, and the amplification curve had obvious exponential growth period.

- (2) The blank control FAM channel had no amplification curve, or the amplification curve was slightly oblique without significant exponential growth, and the Ct value of FAM channel was ≥24.
- (3) Result determination: After determining Ct value and △Ct value according to the above steps, determine the result according to the following table.

Table 2 Result determination

| Mutation<br>type | Negative | Negative | | Positive | |
|---|---|---|---|---|---|
| C2201 | There was no obvious amplification of FAM channels Or the Ct value is not displayed | Ct value < 25 | $\triangle$ Ct > 9 | Ct<br>value <<br>25 | △Ct ≤ 9 |
| C2301 | There was no obvious amplification of FAM channels Or the Ct value is not displayed | Ct value < 25 | $\triangle$ Ct > 9 | Ct<br>value <<br>25 | △Ct ≤ 9 |

#### 4.2 Evaluation method for nucleic acid sequence determination

- (1) The results of the positive reference substance tested on the machine for nucleic acid sequence determination were positive, and the results of the blank reference substance should be in line with expectations without mutation detection.
- (2) Determination of reagent results: the sequencing software Mutation Surveyor was used to interpret the results. When 6695 G>GA, corresponding mutation is indicated; otherwise, no mutation is indicated.

#### 4.3 Evaluate the conformity between the kit and the reference method

- (1) If the results to be tested and the reference results are both positive or negative, it is regarded as in conformity.
- (2) In the event that the result to be tested is positive and the reference result is negative, or the result to be tested is negative and the reference result is positive, it is recorded as nonconformity.

- (3) If the result to be tested fails and the reference method has confirmed results, it shall be recorded as non-conformity. The reasons and results of the non-conformity shall be truthfully recorded, and the comparison results shall be repeatedly confirmed when necessary.
- (4) Complete subsequent statistical analysis based on the above statistical results.

#### 5 Statistical methods

Statistical analysis of clinical study data: Kappa test was used for statistical analysis of the comparison between the kit test results and gene sequencing test results, and then the difference between the results obtained by the two methods was compared. If Kappa > 0.6, it was proved that there was no statistical difference between the two methods in detecting TERT gene promoter mutations in glioma samples.

#### 6 Duration of clinical trials and its reasons

The clinical study lasted about 6-8 months from the drafting of the protocol, project approval, ethical review, agreement signing, specimen collection, the beginning of the test to the end of the trial, and the report and seal are completed. If the sample collection is smooth and the number of samples meets the test requirements, the clinical trial time can be shortened; if it is not smooth, the time can be appropriately extended.

# 7 Inclusion criteria, exclusion criteria and rejection Criteria

#### 7.1 Inclusion criteria

- (1) Be able to provide samples timely according to the requirements of the protocol.
- (2) The pathological examination conforms to the type of tissue sample listed in Table 1, and the tumor content is not less than 50%.
- (3) The sample should have corresponding basic clinical information, including: the patient's visiting No. / medical record No./specimen No., age, sex, and pathological diagnosis result.

#### 7.2 Exclusion criteria

Those who do not meet any of the above conditions are excluded.

Rationale: Included glioma, other brain tumors, and normal samples should be statistically significant and the conclusions obtained are scientifically valid. The selection of subjects for this

study, while excluding research-related influencing factors, has no adverse effect on the health of the subjects.

#### 7.3 Rejection Criteria

- (1) Samples considered by the researcher to be unsuitable for continuing clinical trials, such as samples that have not been prepared in accordance with the required steps.
- (2) Samples with unqualified genomic DNA quality, such as:
  - ① DNA concentration is less than 10ng/μL;
  - ② Genomic DNA was severely degraded or had insufficient purity, and OD260/OD280 exceeded the range of 1.6~2.0.
- (3) Samples whose repeated test results of reference methods failed.
- (4) Samples with incomplete clinical basic information (patients' visiting No. / medical record No./specimen No., age, sex, pathological diagnosis result).

# 8 Provisions for amendments to clinical trial protocols

Any modification to the protocol during the test should be explained, and the time, reason, process and record of the modification should be elaborated in detail, and its impact on the evaluation of the whole study results should be demonstrated.

# 9 Ethical issues and explanations of clinical trials

This clinical trial verification test uses the patient's pathological specimens in the previous treatment process. It is limited to in vitro diagnosis, does not directly contact the patient, does not cause any harm to the patient, and only compares the performance of the reagent with the control reagent. The results are only used for study and analysis related to this test, and will not guide the diagnosis and treatment of patients based on this, so it will not have any adverse effects on the human body. This clinical trial strictly complies with the "Declaration of Helsinki", and this clinical verification trial involves relevant patient data. Such as: Patient visiting No. / medical record No. / specimen No., age, sex, pathological diagnosis result, etc. The hospital and Genetron Health (Beijing) Co., Ltd. will jointly undertake the confidentiality of the patient information, and the clinical trial

operator and clinical validation unit promise not to disclose the content related to the subject specimen.

Therefore, the clinical trial was verified to submit an informed consent exemption to the ETHICS Committee.

# 10 Data processing and record keeping

It is required to keep all experimental records during the clinical trial, the results should be objective, timely and serious, and the operator and operation time should be recorded. Medical institutions shall keep the clinical trial data for five years after the termination of the trial.